CLINICAL TRIAL: NCT06714032
Title: Integrated Traditional Chinese and Conventional Medicine in Treatment for Patients with Severe COVID-19: Study Protocol for a Randomized Controlled Trial
Brief Title: Effect of Traditional Chinese Medicine of Severe COVID-19
Acronym: COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Henan University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TCM for Severe COVID-19
Record Dates: First submitted 2024-10-26; First posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-12

CONDITIONS: Severe COVID-19
Keywords: Traditional Chinese Medicine; Severe COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TCM plus conventional drug (Experimental): The experimental group will receive three type of TCM inaddition conventional drug
  Interventions: Drug: TCM plus conventional drug
- TCM placebo plus conventional drug (Placebo Comparator): The control group will receive three type of placebo TCM inaddition conventional drug
  Interventions: Drug: TCM placebo plus conventional drug

INTERVENTIONS:
Drug: TCM plus conventional drug — All patients were treated according to international guidelines. The Experimental group will receive TCM according to the TCM syndrome.
  Arms: TCM plus conventional drug
Drug: TCM placebo plus conventional drug — All patients were treated according to international guidelines. The control group will receive TCM placebo according to the TCM syndrome.
  Arms: TCM placebo plus conventional drug

SUMMARY:
This study evaluated the effect of integrated traditional Chinese and Western medicine in the treatment of Severe COVID-19. The patients were randomly divided into experimental group and control group.

DETAILED DESCRIPTION:
In this study, a multi center randomized controlled trial design was adopted, and the subjects were randomly divided into the experimental group and the control group. The control group was treated with western medicine conventional treatment plus traditional Chinese medicine decoction simulant, while the experimental group was treated with traditional Chinese medicine syndrome differentiation treatment decoction. The course of treatment was 14 days and the patients were followed up for 3 months. The clinical effect of integrated traditional Chinese and Western medicine treatment was evaluated from the aspects of 28 day mortality, 28 days without invasive mechanical ventilation, invasive mechanical ventilation rate, 28 days without ICU stay, clinical stability time, length of hospital stay, quality of life, SOFA score, etc., to clarify the clinical efficacy of integrated traditional Chinese and Western medicine treatment for Severe COVID-19 infection.

ELIGIBILITY:
Inclusion Criteria:

* accord with the diagnosis of severe/critical novel coronavirus infection;
* Age > 18 years old;
* TCM syndrome differentiation diagnosis by the attending physician or above or two attending physicians for diagnosis and consensus;
* Sign the informed consent form.

Exclusion Criteria:

* Pregnant and lactating women;
* Trauma, hematological malignancies, various solid tumors and obstetric complications;
* Dementia, various mental patients and those who are unwilling to cooperate;
* The patient is expected to die within the next 24 hours;
* Combined with neuromuscular diseases affecting respiratory and motor functions;
* people who have been bedridden for a long time for various reasons;
* Clinical trial participants who are taking part in other intervention measures;
* Those who are known to be allergic to the therapeutic drugs in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2023-01-29 (Actual); Primary Completion 2023-11-08 (Actual); Study Completion 2024-01-25 (Actual)

PRIMARY OUTCOMES:
28-day mortality | Mortality on the 28th day of treatment
  Proportion of patients who died of disease on day 28

SECONDARY OUTCOMES:
Days without invasive mechanical ventilation | the 28 days of the treatment phase
  Days without invasive mechanical ventilation in 28 days
invasive mechanical ventilation rate | 28 days in the treatment phase
  Rate of patients receiving invasive mechanical ventilation
days of non-ICU | 28 days in the treatment phase
  Calculate the number of days of patients not staying in ICU within 28 days
time to clinical stability | every day in the treatment.
  temperature of 37.2°C orlower, heart rate of 100 beats/min or lower, systolic blood pressure of 90 mm Hg or higher, and arterial oxygen tension of 60 mm Hg or higher when the patient was not receiving supplemental oxygen.
hospitalization time | the 28 days of the treatment phase
  length of hospital stays will be recorded.
Clinical status of patients 15 days after randomization | The clinical status of patients was observed 15 days after randomization.
  According to the 6-point clinical improvement scale of the World Health Organization, the lowest score was 1 and the highest was 6. The higher the score, the worse the result.
Quality of life | The scores on the 1st, 4th, 7th, 14th, 21st and 28th day of admission were counted.
  Score according to the quality of life table,the minimum score is 12 points, and the maximum score is 60 points. The higher the score, the worse the result.
TCM syndrome score | The scores on the 1st, 4th, 7th, 14th, 21st and 28th day of admission were counted.
  Traditional Chinese Medicine Syndrome Points.Including cough, expectoration, dyspnea, chest pain, anorexia and fatigue, each item is rated as 1-5 points from mild to severe.The minimum score is 6 points and the maximum score is 30 points. The higher the score, the worse the result.
SOFA score | The scores on the 1st, 4th, 7th, 14th, 21st and 28th day of admission were counted
  Sequential Organ Failure Assessment.It is a scoring system for evaluating and monitoring the organ function of critically ill patients.The minimum score is 0 and the maximum is 24. The higher the score, the worse the result.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Henan University of Traditional Chinese Medicine, Zhengzhou, Henan, China